CLINICAL TRIAL: NCT00358800
Title: A Randomized Cross Over Study to Compare REMStar Auto With C-Flex to Standard CPAP Therapy in Patients With OSAHS, and to Assess Its Safety, Tolerability and Efficacy and Preference Over CPAP.
Brief Title: REMStar Auto With C-Flex - In-Laboratory Performance v. Conventionally Titrated CPAP Therapy: Performances and Preferences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C04-0474
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2006-08-01 (Estimated); Status verified 2006-07

CONDITIONS: Obstructive Sleep Apnoea Hypopnoea Syndrome
Keywords: OSAHS and REMStar Auto with C-Flex
MeSH Terms: conditions — Sleep Apnea, Obstructive

INTERVENTIONS:
Device: REMStar Auto with C-Flex

SUMMARY:
This study will evaluate the use of REMStar Auto with C-Flex (RSA C-Flex) therapy in subjects with previously diagnosed obstructive sleep apnea / hypopnea syndrome, during in-laboratory studies. The study will determine the ability of RSA C-Flex therapy to effectively treat the sleep apnea events. Mask leak and key sleep parameters will be monitored, and are expected to be improved with C-Flex vs. CPAP therapy. Satisfaction from both patient and technician will also be monitored.

DETAILED DESCRIPTION:
The research question we are exploring is whether the To determine if treatment with C-FLEX is at least equivalent to conventional CPAP therapy as evidenced by standard sleep and breathing variables and To determine if the treatment with C-FLEX has a positive impact as determined by patient and technologist assessment of the PSG experience.

Sleep laboratory rooms will be configured with a RSA device, which can deliver either conventional CPAP or Auto CPAP with C-Flex. Each night the subjects eligible for the trial will be interviewed, and consented for the study. The subjects will be instrumented for polysomnography and PAP titration (with PSG recording of RSA flow, estimated tidal volume, pressure, and estimated leak - via the Analog Output Module). Each subject will be instructed in PAP therapy (using standard methods), and have an appropriate patient interface selected per standard laboratory protocol. Each night, the patients will be randomized to either therapy (conventional CPAP therapy without C-Flex, or RSA C-Flex). PSG will be schedules to take place on consecutive nights when possible. The patient will not be aware of the therapy they will be subjected to, but the night technician will be aware of the therapy choice. On the next night, the subject will receive the alternative therapy (cross-over).

Conventional CPAP without C-Flex CPAP pressure will be set to the therapy pressure determined during a previous titration study. Technicians will record all interactions with the subject, as well as any equipment used in the study. Study data will be analyzed for standard polysomnographic outcome parameters listed below. Patient will complete a visual analog satisfaction questionnaire following the study.

RSA with C-Flex RSA C-Flex will be set with pressure range from 4 to 20 cmH2O. Patients will be arbitrarily set to a C-Flex comfort setting of 3 (maximum pressure relief). If the patient comments about any sensation of 'breathlessness' due to the pressure relief, comfort setting may be adjusted to 2 or 1 by the night technician. The subject is not informed of the therapy selected for the study. Technicians will record all interactions with the subject, as well as any equipment used in the study. Study data will be analyzed for standard polysomnographic outcome parameters listed below. Patient will complete a visual analog satisfaction questionnaire following the study.

Demographic Data: Age, gender composition, body mass index, and baseline (diagnostic) AHI will be presented with descriptive statistics. Appropriate statistical analysis will be performed to compare the results of the titration night with REMStar Auto to the night on conventional CPAP. Laboratory Experience: Number of interactions, types of interactions, equipment used and VAS of both patient and technician will be recorded for each subject. Polysomnographic Data, Cardiopulmonary and the process data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Primary medical diagnosis Obstructive Sleep Apnea / Hypopnea Syndrome
* AHI ≥ 15 events•hr-1 of sleep
* Ability to provide consent
* Successful completion of a conventional CPAP titration in a sleep laboratory under polysomnographic conditions (success defined by reduction of AHI to < 5•hr-1 during therapeutic portion of study, in supine position and in REM and NREM sleep state).

Exclusion Criteria:

* Patients who are medically complicated or who are medically unstable.
* Patients who have been on chronic CPAP or BiPAP therapy or require oxygen therapy.
* Patients with respiratory failure or respiratory insufficiency or who have elevated arterial carbon dioxide levels while awake.
* Patients who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days.
* Patients with non-OSA sleep disorders.
* Patients in whom PAP therapy is otherwise medically contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-02; Study Completion 2005-12

PRIMARY OUTCOMES:
This study will compare apnea-hypopnea index (AHI) and standard sleep and breathing variables while on nasal CPAP vs REMStar Auto with C-Flex. Subject himself acts his own control

SECONDARY OUTCOMES:
The study will also compare Polysomnographic Data.
This study will compare Cardiopulmonary
This study will compare Technician interactions with subject

CONTACTS AND LOCATIONS:
Overall Officials: Najib Ayas, Principal Investigator — The University of British Columbia
Locations (1):
- UBC Sleep Disorder Program and Sleep Lab, UBC Hospital, Vancouver, British Columbia, Canada